CLINICAL TRIAL: NCT01259089
Title: A Phase I/II Trial of Hsp 90 Inhibitor AUY-922 in Patients With Lung Adenocarcinoma With "Acquired Resistance" to EGFR Tyrosine Kinase Inhibitors
Brief Title: Hsp90 Inhibitor AUY922 and Erlotinib Hydrochloride in Treating Patients With Stage IIIB-IV Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Robert H. Lurie Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 10L01; STU00038215 (Other: Northwestern University IRB)
Record Dates: First submitted 2010-12-10; First posted 2010-12-13 (Estimated); Results first posted 2018-11-21 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2018-10

CONDITIONS: Adenocarcinoma of the Lung; Non-small Cell Lung Cancer
Keywords: Adenocarcinoma of the Lung; Non-small Cell Lung Cancer
MeSH Terms: conditions — Adenocarcinoma of Lung; Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; 5-(2,4-dihydroxy-5-isopropylphenyl)-4-(4-morpholin-4-ylmethylphenyl)isoxazole-3-carboxylic acid ethylamide; Biopsy, Needle

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients receive Hsp90 inhibitor AUY922 IV over 1 hour once weekly and oral erlotinib hydrochloride once daily. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: erlotinib hydrochloride; Drug: Hsp90 inhibitor AUY922; Other: laboratory biomarker analysis; Procedure: needle biopsy; Genetic: mutation analysis; Other: pharmacological study

INTERVENTIONS:
Drug: erlotinib hydrochloride — Given orally
  Other Names: CP-358,774; erlotinib; OSI-774; Tarceva
Drug: Hsp90 inhibitor AUY922 — Given IV
  Other Names: AUY922
Other: laboratory biomarker analysis — Correlative studies
Procedure: needle biopsy — Undergo image-guided needle biopsy (correlative studies)
  Other Names: aspiration biopsy; puncture biopsy
Genetic: mutation analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
Hsp90 inhibitor AUY922 and erlotinib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. This phase I/II trial is studying the side effects and best dose of Hsp90 inhibitor AUY922 when given together with erlotinib hydrochloride and to see how well it works in treating patients with stage IIIB-IV non-small cell lung cancer.

DETAILED DESCRIPTION:
This is a phase I, dose-escalation study of Hsp90 inhibitor AUY922 followed by a phase II study. Patients receive Hsp90 inhibitor AUY922 IV over 1 hour once weekly and oral erlotinib hydrochloride once daily. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity. After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have pathologic evidence of advanced lung adenocarcinoma (stage IIIB or stage IV) confirmed histologically/cytologically at NU, MSKCC, or DFCI and EITHER previous RECIST-defined response (CR or PR) to an EGFR-TKI (erlotinib or gefitinib) or an investigational EGFR TK inhibitor OR a documented mutation in the EGFR gene (G719X, exon 19 deletion, L858R, L861Q)
* Radiographic progression by RECIST during treatment with erlotinib/gefitinib
* Received treatment with erlotinib/gefitinib throughout the one month prior to enrollment and at least six months at any time
* Measurable (RECIST) indicator lesion not previously irradiated
* Must have undergone a biopsy after the development of acquired resistance
* Karnofsky Performance Status >= 70% OR ECOG/WHO Performance Status 0-1
* Signed informed consent
* Effective contraception and negative serum pregnancy test obtained within two weeks prior to the first administration of AUY922 in all pre-menopausal women (ie., last menstrual period =< 24 months ago) and women < 2 years after onset of menopause; menopause is defined as the time at which fertility ceases, where a woman has had no menstruation for > 24 months
* Total bilirubin =< 1.5 x Upper Limit of Normal (ULN)
* AST/SGOT and ALT/SGPT =< 3.0 x ULN, or =< 5.0 x ULN if liver metastasis present
* Absolute neutrophil count (ANC) >= 1.5 x10^9/L
* Hemoglobin (Hgb) >= 9g/dL
* Platelets (plts) >= 100 x 10^9/L
* Serum creatinine =< 1.5 x ULN or 24 hour clearance >= 50 mL/min

Exclusion Criteria:

* Symptomatic CNS metastases which are symptomatic and /or requiring escalating doses of steroids
* Prior treatment with any HSP90 inhibitor compounds
* Conventional chemotherapy, radiation or monoclonal antibodies within 4 weeks (erlotinib/gefitinib therapy within the past 4 weeks IS allowed)
* Palliative radiation within 2 weeks
* Unresolved diarrhea >= CTCAE grade 2
* Pregnant or lactating women
* Women of childbearing potential (WCBP) (i.e. women able to become pregnant) not using double-barrier methods of contraception (abstinence, oral contraceptives, intrauterine device or barrier method of contraception in conjunction with spermicidal jelly, or surgically sterile); male patients whose partners are WCBP not using double-barrier methods of contraception
* Acute or chronic liver or renal disease
* Other concurrent severe and/or uncontrolled medical conditions that could cause unacceptable safety risks or compromise compliance with the protocol
* Major surgery =< 2 weeks prior to randomization or who have not recovered from such therapy
* History (or family history) of long QT syndrome
* Mean QTc >= 450 msec on baseline ECG
* History of clinically manifested ischemic heart disease =< 6 months prior to study start
* History of heart failure or left ventricular (LV) dysfunction (LVEF =< 45%) by MUGA or ECG
* Clinically significant resting bradycardia (< 50 beats per minute)
* Clinically significant ECG abnormalities including 1 or more of the following: left bundle branch block (LBBB), right bundle branch block (RBBB) with left anterior hemi-block (LAHB); ST segment elevation or depression > 1mm, or 2nd (Mobitz II), or 3rd degree AV block
* History ventricular tachycardia
* Other clinically significant heart disease including congestive heart failure (New York Heart Association class III/IV) or uncontrolled hypertension (> 160/90 despite intensive medical management)
* Patients who are currently receiving treatment with any medication which has a relative risk of prolonging the QTcF interval and cannot be switched or discontinued to an alternative drug prior to commencing AUY922
* Known diagnosis of HIV infection (HIV testing is not mandatory)
* Patients with a history of another primary malignancy that is currently clinically significant or currently requires active intervention
* Patients who are receiving warfarin (Coumadin®) will be excluded unless =< 2 mg/d, with an INR < 1.5
* Patients with known disorders due to a deficiency in bilirubin glucuronidation (e.g. Gilbert's syndrome)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2011-04-27 (Actual); Primary Completion 2013-06-04 (Actual); Study Completion 2014-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Johnson, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Northwestern University, Chicago, Illinois
  - Memorial Sloan-Kettering Cancer Center, New York, New York

REFERENCES:
- [Derived] Johnson ML, Yu HA, Hart EM, Weitner BB, Rademaker AW, Patel JD, Kris MG, Riely GJ. Phase I/II Study of HSP90 Inhibitor AUY922 and Erlotinib for EGFR-Mutant Lung Cancer With Acquired Resistance to Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitors. J Clin Oncol. 2015 May 20;33(15):1666-73. doi: 10.1200/JCO.2014.59.7328. Epub 2015 Apr 13. PMID 25870087

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened for accrual on March 28, 2011 with an accrual goal of up to 30 patients in phase I and 25 patients in phase II. 18 patients were enrolled treated in phase I and 19 patients treated in phase II. The study was closed permanently on May 6, 2013.
Groups:
- Cohort 1 - 25 mg/m2 AUY922+75 mg Daily Erlotinib; Cohort 3 - 37.5 mg/m2 AUY922+150 mg Daily Erlotinib; Cohort 4 - 55 mg/m2 AUY922+150 mg Daily Erlotinib; Cohort 5 - 70 mg/m2 AUY922+150 mg Daily Erlotinib; Phase II- 70 mg/m2 AUY922+150 mg Daily Erlotinib: Patients receive Hsp90 inhibitor AUY922 IV over 1 hour once weekly and 75mg oral erlotinib hydrochloride once daily. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  erlotinib hydrochloride: Given orally
  Hsp90 inhibitor AUY922: Given IV
  laboratory biomarker analysis: Correlative studies
  needle biopsy: Undergo image-guided needle biopsy (correlative studies)
  mutation analysis: Correlative studies
  pharmacological study: Correlative studies
- Cohort 2 - 25 mg/m2AUY922+150 mg Daily Erlotinib: Patients receive Hsp90 inhibitor AUY922 IV over 1 hour once weekly and oral erlotinib hydrochloride once daily. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  erlotinib hydrochloride: Given orally
  Hsp90 inhibitor AUY922: Given IV
  laboratory biomarker analysis: Correlative studies
  needle biopsy: Undergo image-guided needle biopsy (correlative studies)
  mutation analysis: Correlative studies
  pharmacological study: Correlative studies
Period: Reached First Response at 4 Weeks
Arm/Group | Cohort 1 - 25 mg/m2 AUY922+75 mg Daily Erlotinib | Cohort 2 - 25 mg/m2AUY922+150 mg Daily Erlotinib | Cohort 3 - 37.5 mg/m2 AUY922+150 mg Daily Erlotinib | Cohort 4 - 55 mg/m2 AUY922+150 mg Daily Erlotinib | Cohort 5 - 70 mg/m2 AUY922+150 mg Daily Erlotinib | Phase II- 70 mg/m2 AUY922+150 mg Daily Erlotinib
Started | 3 | 3 | 3 | 3 | 6 | 20
Started Treatment on Study | 3 | 3 | 3 | 3 | 6 | 19
Completed 4 Weeks of Treatment | 3 | 3 | 3 | 3 | 6 | 18
Completed | 3 | 3 | 3 | 3 | 6 | 18
Not Completed | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Patient not treated on study | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1
Period: Confirmed Response at 8 Weeks
Arm/Group | Cohort 1 - 25 mg/m2 AUY922+75 mg Daily Erlotinib | Cohort 2 - 25 mg/m2AUY922+150 mg Daily Erlotinib | Cohort 3 - 37.5 mg/m2 AUY922+150 mg Daily Erlotinib | Cohort 4 - 55 mg/m2 AUY922+150 mg Daily Erlotinib | Cohort 5 - 70 mg/m2 AUY922+150 mg Daily Erlotinib | Phase II- 70 mg/m2 AUY922+150 mg Daily Erlotinib
Started | 3 | 3 | 3 | 3 | 6 | 18
Completed | 3 | 3 | 2 | 2 | 2 | 8
Not Completed | 0 | 0 | 1 | 1 | 4 | 10
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 2
Not completed — Progressive disease | 0 | 0 | 1 | 1 | 3 | 7
Period: Continued Treatment After 8 Weeks
Arm/Group | Cohort 1 - 25 mg/m2 AUY922+75 mg Daily Erlotinib | Cohort 2 - 25 mg/m2AUY922+150 mg Daily Erlotinib | Cohort 3 - 37.5 mg/m2 AUY922+150 mg Daily Erlotinib | Cohort 4 - 55 mg/m2 AUY922+150 mg Daily Erlotinib | Cohort 5 - 70 mg/m2 AUY922+150 mg Daily Erlotinib | Phase II- 70 mg/m2 AUY922+150 mg Daily Erlotinib
Started | 3 | 3 | 2 | 2 | 2 | 8
Completed | 1 | 2 | 1 | 1 | 0 | 7
Not Completed | 2 | 1 | 1 | 1 | 2 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 2 | 1
Not completed — Progressive disease | 1 | 1 | 1 | 1 | 0 | 0
Period: Survival Follow up for Two Years
Arm/Group | Cohort 1 - 25 mg/m2 AUY922+75 mg Daily Erlotinib | Cohort 2 - 25 mg/m2AUY922+150 mg Daily Erlotinib | Cohort 3 - 37.5 mg/m2 AUY922+150 mg Daily Erlotinib | Cohort 4 - 55 mg/m2 AUY922+150 mg Daily Erlotinib | Cohort 5 - 70 mg/m2 AUY922+150 mg Daily Erlotinib | Phase II- 70 mg/m2 AUY922+150 mg Daily Erlotinib
Started (All patients that are treated on study go into follow up once they finish treatment.) | 3 | 3 | 3 | 3 | 6 | 19
Completed | 0 | 1 | 1 | 0 | 0 | 0
Not Completed | 3 | 2 | 2 | 3 | 6 | 19
Not completed — Death | 3 | 2 | 2 | 3 | 6 | 13
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 2
Not completed — stopped being followed as study closed | 0 | 0 | 0 | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Arm/Group | Arm I
Number analyzed (Participants) | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 37
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 11
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 4
  White | 21
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 38

OUTCOME MEASURES:

1. Primary Outcome: Maximally Tolerated Dose (MTD) of AUY922 and Erlotinib Treatment Combination (Phase I)
Description: To determine the maximally tolerated dose (MTD), and recommended phase II dose of AUY922 when given in combination with erlotinib for patients with acquired resistance to erlotinib. (Phase I)
  Escalation of dose will be in a 3+3 design. If no dose limiting toxicities (DLTs) are seen in 3 patients enrolled at that dose level, then dose will be escalated to the next dose level and the next 3 patients will be enrolled at that dose. Alternatively, if 1 DLT is seen in 3 patients at that dose level, 3 more patients will be added at that same dose level. If 1 DLT is seen in 6 patients at that dose level, MTD will be determined to be at that dose. If more than 1 DLT is seen at that dose level, then the prior lower dose level will be the considered the MTD.
  DLT is defined as any of the following related to the investigational agent: Death and grade 3 and 4 specific hematological and non-hematological toxicities defined in the protocol.
Time Frame: During the first 4 weeks of treatment for each patient.
Measure: Number; unit: Number of DLTs seen
Groups:
- Cohort 1 - 25 mg/m2 AUY922+75 mg Daily Erlotinib; Cohort 2 - 25 mg/m2AUY922+150 mg Daily Erlotinib; Cohort 3 - 37.5 mg/m2 AUY922+150 mg Daily Erlotinib; Cohort 4 - 55 mg/m2 AUY922+150 mg Daily Erlotinib; Cohort 5 - 70 mg/m2 AUY922+150 mg Daily Erlotinib: Patients receive Hsp90 inhibitor AUY922 IV over 1 hour once weekly and oral erlotinib hydrochloride once daily. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  erlotinib hydrochloride: Given orally
  Hsp90 inhibitor AUY922: Given IV
  laboratory biomarker analysis: Correlative studies
  needle biopsy: Undergo image-guided needle biopsy (correlative studies)
  mutation analysis: Correlative studies
  pharmacological study: Correlative studies
Arm/Group | Cohort 1 - 25 mg/m2 AUY922+75 mg Daily Erlotinib | Cohort 2 - 25 mg/m2AUY922+150 mg Daily Erlotinib | Cohort 3 - 37.5 mg/m2 AUY922+150 mg Daily Erlotinib | Cohort 4 - 55 mg/m2 AUY922+150 mg Daily Erlotinib | Cohort 5 - 70 mg/m2 AUY922+150 mg Daily Erlotinib
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 6
Number of DLTs seen | 0 | 0 | 0 | 0 | 1

2. Primary Outcome: Overall Response Rate (ORR), Defined as Complete Response(CR) + Partial Response (PR) Using the Modified RECIST 1.1 Criteria for All Patients Treated at Dose of 70mg/m2 AUG922
Description: Overall response rate (ORR) will be measured per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT scan or MRI:
  Complete response (CR) defined as disappearance of all target lesions. Partial Response (PR), defined as >=30% decrease in the sum of the longest diameter of target lesions.
  Stable Disease (SD) defined as neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum diameters while on study.
  Progressive Disease (PD) defined as having at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started or the appearance of one or more new lesions
Time Frame: At 8 weeks from treatment initiation
Population: All patients that were treated at the MTD dose of 70mg/m2 AUG922 IV were evaluable for this outcome measure (This includes patients treated in cohort 5 of phase I and all patients treated in phase II of the study)
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I
Number analyzed (Participants) | 25
Participants | 4

3. Secondary Outcome: Toxicity as Assessed by NCI CTCAE Version 4.00 When AUG922 Administered at Its MTD (Phase I and II)
Description: To characterize the toxicity profile for the combination of erlotinib and AUY922.
  Toxicity data will be collected every week for the first 28 day cycle and then every two weeks during treatment and up to 28 days after the last treatment. Adverse events will be graded according to the National Cancer Institute's Common Toxicity Criteria for adverse events version 4.0 (CTCAE v4.0). In general adverse events (AEs) will be graded according to the following:
  Grade 1 Mild AE Grade 2 Moderate AE Grade 3 Severe AE Grade 4 Life-threatening or disabling AE Grade 5 Death related to AE
Time Frame: At weeks 1 through 4 and then every 2 weeks during treatment and 30 days post last treatment for up to 2 years and half years
Population: Toxicity collected from all patients treated at the MTD of 70mg/m2 AUY922. 6 patients in phase I and 19 patients in phase II were treated at this dose.
Measure: Number; unit: participants
Arm/Group | Arm I
Number analyzed (Participants) | 25
participants
  Diarrhea | 24
  Skin rash | 16
  Hyperglycemia | 23
  Night blindness | 18
  Hypoalbuminemia | 21
  Fatigue | 11
  Elevated AST | 17
  Nausea | 9
  Hyponatremia | 17
  Elevated bilirubin | 16
  Elevated ALT | 14
  Myalgias/arthralgias | 9
  Visual complaints | 10
  Vomiting | 8
  Elevated APL | 10
  Decreased leukocytes | 10
  Hypokalemia | 10
  Pruritis/dry skin | 5
  Hypocalcemia | 8
  Anemia | 4
  Mucositis | 6
  Decreased lymphocytes | 6
  Decreased platelets | 6
  Hypomagnesemia | 6
  Decreased neutrophils | 5

4. Secondary Outcome: Incidence of Reported Adverse Events in Phase I
Description: Adverse events will be collected weekly for the first 28 day cycle and then every two weeks during treatment and up to 28 days after the last treatment. Adverse events will be graded according to the National Cancer Institute's Common Toxicity Criteria for adverse events version 4.0 (CTCAE v4.0). In general adverse events (AEs) will be graded according to the following:
  Grade 1 Mild AE Grade 2 Moderate AE Grade 3 Severe AE Grade 4 Life-threatening or disabling AE Grade 5 Death related to AE
Time Frame: At weeks 1 through 4 and then every 2 weeks during treatment and 30 days post last treatment, for up to 2 years and half years
Population: Most frequent adverse events for patients treated with 25 to 55mg/m2 dose of AUY9222.
Measure: Number; unit: participants
Arm/Group | Arm I
Number analyzed (Participants) | 12
participants
  Diarrhea | 11
  Skin rash | 9
  Hyperglycemia | 0
  Night blindness | 3
  Hypoalbuminemia | 0
  Fatigue | 8
  Elevated AST | 1
  Nausea | 8
  Hyponatremia | 0
  Elevated bilirubin | 0
  Elevated ALT | 0
  Myalgias/arthralgias | 5
  Visual complaints | 4
  Vomiting | 4
  Elevated ALP | 0
  Decreased leukocytes | 0
  hypokalemia | 0
  Pruritis/dry skin | 4
  Hypocalcemia | 0
  anemia | 2
  Mucositis | 0
  Decreased lymphocytes | 0
  Decreased platelets | 0
  Hypomagnesemia | 0
  Decreased neutrophils | 0

5. Secondary Outcome: Progression-free Survival (Phase II)
Description: Median Progression Free Survival (PFS) will be calculated from time of treatment initiation until the first documentation of progressive disease. Patients will be considered to have progressive disease when CT scan or MRI show at least a 20% increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: From the time of first treatment with AUY922 to disease progression for up to 2 years post treatment
Population: 25 of the patients were treated at the MTD and were evaluable for progression free survival. Data was collected up until September 30 2014 when study was closed permanently and no further data was collected for patients survival due to IND withdrawal.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm I
Number analyzed (Participants) | 25
Months | 1.7 [1.1 to 4.9]

6. Secondary Outcome: Overall Survival (Phase II)
Description: Overall survival (OS) is defined as the time from treatment initiation until death due to any cause.
Time Frame: From the time of first treatment with AUY922 to death, followed up to 2 years post treatment
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm I
Number analyzed (Participants) | 25
Months | 7.4 [4.0 to 17.9]

7. Secondary Outcome: Overall Survival Among Patients With Acquired Resistance With T790M Mutations (Phase II)
Description: Overall Survival (OS) will be measured from treatment initiation until death due to any cause for patients with acquired resistance with T790M mutations in the phase II portion of the study.
Time Frame: From the time of first treatment with AUY922 to death, followed for up to 2 years
Population: No data was collected or analyzed for this outcome measure. There is no data to report. IND was withdrawn before the studies anticipated termination date.
Arm/Group | Arm I
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected weekly for the first 28 day cycle and then every two weeks up to 2 and half year period.
Description: Only highest grade lab AEs were collected for each patient. All other AEs were collected as defined by clinicaltrials.gov. Phase I+II data collected together as toxicity objectives for the study were looking at AEs in relation to this combination of treatment rather than treatment dose.
Arm/Group | Cohort 1 - 25 mg/m2 AUY922+75 mg Daily Erlotinib | Cohort 2 - 25 mg/m2AUY922+150 mg Daily Erlotinib | Cohort 3 - 37.5 mg/m2 AUY922+150 mg Daily Erlotinib | Cohort 4 - 55 mg/m2 AUY922+150 mg Daily Erlotinib | Cohort 5 - 70 mg/m2 AUY922+150 mg Daily Erlotinib | Phase II- 70 mg/m2 AUY922+150 mg Daily Erlotinib
All-Cause Mortality (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 3/3 | 6/6 | 13/19
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/3 | 1/3 | 1/3 | 2/6 | 1/19
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 3/3 | 6/6 | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 - 25 mg/m2 AUY922+75 mg Daily Erlotinib (N=3) | Cohort 2 - 25 mg/m2AUY922+150 mg Daily Erlotinib (N=3) | Cohort 3 - 37.5 mg/m2 AUY922+150 mg Daily Erlotinib (N=3) | Cohort 4 - 55 mg/m2 AUY922+150 mg Daily Erlotinib (N=3) | Cohort 5 - 70 mg/m2 AUY922+150 mg Daily Erlotinib (N=6) | Phase II- 70 mg/m2 AUY922+150 mg Daily Erlotinib (N=19)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Patient also experienced anemia
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Patient also experienced diarrhea and anemia
Ileal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Patient also had seizure due to not being able to take keppa because of nausea and vomiting.
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumor pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2)
Conduction disorder (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Progressive disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Worsening symptoms included dyspnea and pleural effusion
Diarrhea with blood (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 - 25 mg/m2 AUY922+75 mg Daily Erlotinib (N=3) | Cohort 2 - 25 mg/m2AUY922+150 mg Daily Erlotinib (N=3) | Cohort 3 - 37.5 mg/m2 AUY922+150 mg Daily Erlotinib (N=3) | Cohort 4 - 55 mg/m2 AUY922+150 mg Daily Erlotinib (N=3) | Cohort 5 - 70 mg/m2 AUY922+150 mg Daily Erlotinib (N=6) | Phase II- 70 mg/m2 AUY922+150 mg Daily Erlotinib (N=19)
Anemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 1 | 3
Atrioventricular block first degree (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Chest pain (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Titnnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1
Blurred vision (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 3
Cataract (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Corneal ulcer (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Flashing lights (Eye disorders) | 0 | 1 | 0 | 1 | 1 | 0
Floaters (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1
Night blindness (Eye disorders) | 0 | 1 | 0 | 2 | 4 | 14
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 2 | 3 | 3
Diarrhea (Gastrointestinal disorders) | 3 | 3 | 3 | 2 | 5 | 19
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 5
Nausea (Gastrointestinal disorders) | 2 | 2 | 3 | 1 | 2 | 7
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 0 | 8
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 3 | 3 | 3 | 3 | 5 | 18
Fever (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 2 | 0 | 0 | 0 | 1 | 1
Eye Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Mucosal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Papulopustular rash (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
Paronychia (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 2
Upper Respiratory Infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 4 | 10
Alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 9
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 1 | 16
Cholesterol high (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 3
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 2 | 4
Weight loss (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
White blood cell decreased (Investigations) | 0 | 0 | 0 | 0 | 2 | 8
Blood Bilirubin Increased (Investigations) | 0 | 0 | 0 | 0 | 3 | 13
Activated Partial Thromboplastin time Prolonged (Investigations) | 0 | 0 | 0 | 0 | 1 | 3
INR Increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 1
Platelet Count Decreased (Investigations) | 0 | 0 | 0 | 0 | 2 | 4
Neutrophil Count Decreased (Investigations) | 0 | 0 | 0 | 0 | 2 | 3
Serum Amylase Increased (Investigations) | 0 | 0 | 0 | 0 | 3 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 4 | 18
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 5 | 16
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 6
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 8
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 5
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 3 | 14
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 3
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypernatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Joint Range of Motion Decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Muscle Weakness, Left-sided (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Muscle Weakness Lower Limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1
Paresthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 | 0 | 1 | 1 | 3 | 9
Seizure (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 2 | 3 | 6 | 16
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 3 | 5 | 12
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1 | 2 | 1
Erythema Multiforme (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hirsutism (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 2 | 3
Rash Acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 3 | 4
Rash Maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 1 | 1 | 4
Menopause (Social circumstances) | 0 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 4
Thromboembolic event (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Bleeding (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Bleeding gums (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Blood in sputum (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Visual Disturbances (Eye disorders) | 0 | 0 | 0 | 0 | 2 | 3
Trichiasis of the eyelid (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Fissures (General disorders) | 0 | 0 | 0 | 1 | 0 | 2
Clostridium Difficile (C Diff) (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Decreased Appetite (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cold intolerance (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Taste changes (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Bruise at port site (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Night Sweats (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Reaction at port site (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Muscle cramps (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 4
Tremors (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Leg and hip pain/weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Rash from cut (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Sores in mouth (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Redness on bottom lip (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
New progressive leptomeningeal disease (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Data was collected up until September 30 2014 when study was closed permanently and no further data was collected for patients survival due to IND withdrawal.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No